CLINICAL TRIAL: NCT02405507
Title: The Effect of Wheat Germ on Gastrointestinal Discomfort, Blood Cholesterol and Postprandial Glycaemic Response in Healthy Volunteers
Brief Title: The Effect of Wheat Germ on Gastrointestinal Discomfort, Blood Cholesterol and Postprandial Glycaemic Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Center for Health Technology and Services Research (Other); Project VALORINTEGRADOR financed by COMPETE (FCOMP-01-0202-FEDER-038861) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: VI001
Record Dates: First submitted 2015-03-11; First posted 2015-04-01 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers
Keywords: Gastrointestinal Discomfort; Wheat germ; Constipation; Glycaemic Index; Blood Cholesterol Level; Glycaemic Response; Cholesterol; PAC-SYM; Gut Microbiota
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- wheat bread with wheat germ (Experimental): wheat bread with wheat germ supplementation
  Interventions: Dietary Supplement: wheat bread with wheat germ
- wheat bread without wheat germ (Placebo Comparator): wheat bread without wheat germ supplementation
  Interventions: Dietary Supplement: wheat bread without wheat germ

INTERVENTIONS:
Dietary Supplement: wheat bread with wheat germ
  Arms: wheat bread with wheat germ
Dietary Supplement: wheat bread without wheat germ
  Arms: wheat bread without wheat germ

SUMMARY:
Wheat germ is a by-product of the wheat-milling industry with high nutritional value and therefore could be used as a raw source for the preparation of food products such as bread, cookies, muffins, etc.

The aim of this study is to assess the effects of ingesting wheat breads supplemented with wheat germ on gastrointestinal discomfort, blood cholesterol and postprandial glycaemic response in healthy human volunteers.

DETAILED DESCRIPTION:
This is a crossover, double blinded, placebo controlled randomized trial. The study will compare the effect of consumption of wheat breads with or without wheat germ on healthy individuals, during 2 intake periods of 4 weeks each and 5 weeks washout before crossover.

The study will focus on the effects of wheat breads supplemented with wheat germ on gastrointestinal discomfort, blood cholesterol and postprandial glycaemic response in healthy human volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women
* Age 18 - 60 years
* Healthy volunteers free of chronic diseases with relevant effect on the gastrointestinal system or on visceral motility
* Without a diagnosis of any digestive disease including functional bowel disorders such as IBS
* Non-diabetic, no gastric bypass surgery
* Have a fasting plasma glucose (finger-stick) <100 mg/dl (<5.5 mmol/L)
* Non-smoker
* Willing and able to provide written informed consent

Exclusion Criteria:

* Subject under prescription for medication for digestive symptoms such as anti-spasmodic, laxatives and anti-diarrheic drugs or other digestive auxiliaries
* Relevant history, presence of any medical disorder or intake of medication / dietary supplements, potentially interfering with this trial at screening
* Subjects with stool frequency of ≤ 1 stool every 7 days
* Subjects not willing to avoid pre- and probiotics for the duration of the study
* Intake of antibiotics in the last 4 weeks and laxatives in the last 2 weeks
* Current use of medication for lowering blood cholesterol or glucose
* Change of dietary habits within the 4 weeks prior to screening (for instance start of a diet high in fibres)
* Pregnant subject or subject planning to become pregnant during the study; breast-feeding subject
* Subjects with history of drug, alcohol or other substances abuse, or other factors limiting their ability to co-operate during the study
* Participants anticipating a change in their lifestyle or physical activity levels since this may also influence the results
* Known food intolerance or allergy
* Subject involved in any clinical or food study within the preceding month

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Changes in mean Patient Assessment of Constipation Symptoms (PAC-SYM) score from baseline to weeks 2, 4, 7, 9, 11 and 13 | at the end of week 0 (after 2-week run-in period), at the end of weeks 2 and 4 (during 4-week intake period), at the end of weeks 7 and 9 (during 5-week washout period), at the end of weeks 11 and 13 (during 4-week intake period after crossover)
  A validated PAC-SYM questionnaire will be used. PAC-SYM is a 12-item, self-administered questionnaire used to measure severity of symptoms over the past 2 weeks in patients with constipation. The PAC-SYM questionnaire has been demonstrated and documented to have internal consistency, reproducibility, validity, sensitivity, and responsiveness. PAC-SYM items are rated on a 5-point scale (0=absent, 1=mild, 2=moderate, 3=severe, 4=very severe) and grouped into three subscales related to abdominal symptoms (bloating, discomfort, pain, and cramps), stool symptoms (incomplete bowel movement, false alarm, straining, too hard, and too small), and rectal symptoms (painful bowel movement, burning, and bleeding or tearing). The total score and subscale scores are computed by taking the mean of item responses (score range 0-4). A reduction in score reflects an improvement in symptoms. Cultural adaptation and linguistic validation of the PAC-SYM for Portugal was performed by Mapi Research.
Changes in fasting serum total cholesterol from baseline to visit 2, 3 and 4 | at visit 1 (after 2-week run-in period), visit 2 (after 4-week intake period), visit 3 (after 5-week washout period) and visit 4 (after 4-week intake period after crossover)
Changes in fasting serum triglycerides from baseline to visit 2, 3 and 4 | at visit 1 (after 2-week run-in period), visit 2 (after 4-week intake period), visit 3 (after 5-week washout period) and visit 4 (after 4-week intake period after crossover)
Changes in fasting serum high-density lipoprotein (HDL) cholesterol from baseline to visit 2, 3 and 4 | at visit 1 (after 2-week run-in period), visit 2 (after 4-week intake period), visit 3 (after 5-week washout period) and at visit 4 (after 4-week intake period after crossover)
Changes in fasting serum low-density lipoprotein (LDL) cholesterol from baseline to visit 2, 3 and 4 | at visit 1 (after 2-week run-in period), visit 2 (after 4-week intake period), visit 3 (after 5-week washout period) and at visit 4 (after 4-week intake period after crossover)
Changes in fasting serum C-reactive protein from baseline to visit 2, 3 and 4 | at visit 1 (after 2-week run-in period), visit 2 (after 4-week intake period), visit 3 (after 5-week washout period) and at visit 4 (after 4-week intake period after crossover)
Changes in capillary blood glucose from baseline to visit 2 and 4 | 0, 30, 60 and 120 minutes post-meal: at visit 1 (after 2-week run-in period), visit 2 (after 4-week intake period), visit 3 (after 5-week washout period) and at visit 4 (after 4-week intake period after crossover)

SECONDARY OUTCOMES:
Changes in mean Patient Assessment of Constipation Quality of Life (PAC-QOL) score from baseline to weeks 2, 4, 7, 9, 11 and 13 | at the end of week 0 (after 2-week run-in period), at the end of weeks 2 and 4 (during 4-week intake period), at the end of weeks 7 and 9 (during 5-week washout period), at the end of weeks 11 and 13 (during 4-week intake period after crossover)
  A validated PAC-QOL questionnaire will be used. PAC-QOL questionnaire is a 28-item self-administered questionnaire that is being used to measure health-related quality of life (over the past 2 weeks) in patients with chronic constipation. The 28 items are grouped into four subscales: physical discomfort, psychosocial discomfort, worries and concerns, and satisfaction. Previous studies have shown that PAC-QOL is internally consistent, reproducible, valid and responsive to improvements in chronic constipation over time. Cultural adaptation and linguistic validation of the PAC-QOL for Portugal was performed by Mapi Research Trust.
Changes in intestinal microbiota from baseline to visit 2, 3 and 4 | at visit 1 (after 2-week run-in period), visit 2 (after 4-week intake period), visit 3 (after 5-week washout period), and visit 4 (after 4-week intake period after crossover)
Changes in mean daily abdominal discomfort score from baseline to weeks 1, 2, 3, 4, 10, 11, 12 and 13 | daily during run-in period (weeks -1 and 0), intake period (weeks 1, 2, 3, 4, 10, 11, 12 and 13), and washout period (weeks 5, 6, 7, 8 and 9)
  A number scale will be used to measure the average intensity (abdominal discomfort and bloating), over the previous 24 hours, on a 5-point scale from 0 (absence of symptom) to 4 (very severe). Will be assessed through daily records.
Changes in stool consistency from baseline to weeks 1, 2, 3, 4, 10, 11, 12 and 13 | at days with stool during run-in period (weeks -1 and 0), intake period (weeks 1, 2, 3, 4, 10, 11, 12 and 13), and washout period ( weeks 5, 6, 7, 8 and 9)
  The Bristol stool scale will be used to measure the stool consistency. Will be assessed through daily records.
Changes in stool frequency from baseline to weeks 1, 2, 3, 4, 10, 11, 12 and 13 | at days with stool during run-in period (weeks -1 and 0), intake period (weeks 1, 2, 3, 4, 10, 11, 12 and 13), and washout period ( weeks 5, 6, 7, 8 and 9)
  Will be assessed through daily records.
Changes in fasting plasma insulin from baseline to visit 2 and 4 | at visit 1 (after 2-week run-in period), visit 2 (after 4-week intake period), visit 3 (after 5-week washout period) and at visit 4 (after 4-week intake period after crossover)
Changes in mean Perceived Stress Scale (PSS) score from baseline to weeks 4, 9 and 13 | at the end of week 0 (after 2-week run-in period), at the end of week 4 (after 4-week intake period), at the end of week 9 (after 5-week washout period), and at the end of week 13 (after 4-week intake period after crossover)
  A validated Perceived Stress Scale (PSS) self-administered questionnaire with 13-item will be used to measure perceived stress of respondents during the last month (Portuguese version keeps 13 of the 14 original items). The PSS questionnaire has been demonstrated to have internal consistency, reproducibility, validity, and sensitivity. Cultural adaptation and linguistic validation of the PSS for Portugal was implemented by Pais-Ribeiro & Marques (2009).

OTHER OUTCOMES:
Adverse events | at visit 2 (after 4-week intake period), visit 3 (after 5-week washout period), and visit 4 (after 4-week intake period after crossover)
  Registration of any adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Conceição Calhau, PhD, Principal Investigator — CINTESIS, Faculty of Medicine of the University of Porto
Locations (2):
- Portugal (2):
  - PtCRIN, Lisbon
  - CINTESIS - Faculty of Medicine of the University of Porto, Porto

REFERENCES:
- [Result] Moreira-Rosario A, Marques C, Pinheiro H, Norberto S, Sintra D, Teixeira JA, Calhau C, Azevedo LF. Daily intake of wheat germ-enriched bread may promote a healthy gut bacterial microbiota: a randomised controlled trial. Eur J Nutr. 2020 Aug;59(5):1951-1961. doi: 10.1007/s00394-019-02045-x. Epub 2019 Jul 19. PMID 31325040
- [Result] Moreira-Rosario A, Pinheiro H, Marques C, Teixeira JA, Calhau C, Azevedo LF. Does intake of bread supplemented with wheat germ have a preventive role on cardiovascular disease risk markers in healthy volunteers? A randomised, controlled, crossover trial. BMJ Open. 2019 Jan 17;9(1):e023662. doi: 10.1136/bmjopen-2018-023662. PMID 30659039
- [Derived] Moreira-Rosario A, Pinheiro H, Calhau C, Azevedo LF. Can wheat germ have a beneficial effect on human health? A study protocol for a randomised crossover controlled trial to evaluate its health effects. BMJ Open. 2016 Nov 10;6(11):e013098. doi: 10.1136/bmjopen-2016-013098. PMID 28157671